CLINICAL TRIAL: NCT06655649
Title: Impact of Exogenous Ketones on Sleep Disruption in Vulnerable Populations: Phase I Study (KETO-SLEEP 1)
Brief Title: Impact of Exogenous Ketones on Sleep Disruption in Vulnerable Populations
Acronym: KETO-SLEEP 1
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding changes, may resume later in 2025
Sponsor: Johns Hopkins University (Other)
Collaborators: HVMN Inc (Industry); KETONE-IQ (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00439273
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea; Sleep
Keywords: sleep apnea; ketones; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Ketosis | interventions — 1,3-butylene glycol

STUDY DESIGN:
Intervention Model Description: Participants with a history of moderate-severe sleep apnea, who are using CPAP, will be included. KETO-SLEEP 1 (n=20) will examine the pharmacokinetics, GI tolerability, and sleep impacts of ingesting open-label Ketone-IQ (1,3-butanediol) before sleep at 2 doses (20 or 40 g). All sleep studies are performed at home while using CPAP. at home. Some nights will involve ingesting Ketone-IQ before bedtime and wearing a sleep monitoring device (Sleep Profiler). Other nights involve waking up to check capillary ketone levels. Questionnaires will be given to ask about sleep quality and GI tolerability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketone Intervention (Experimental): Participants with sleep apnea using CPAP will undergo open-label procedures. They will ingest (1) nothing, (2) Ketone IQ 20 g or (3) Ketone IQ 40 g before bedtime and undergo objective and subjective sleep assessments.
  Interventions: Dietary Supplement: Ketone-IQ (1,3 Butanediol)

INTERVENTIONS:
Dietary Supplement: Ketone-IQ (1,3 Butanediol) — Ketone-IQ (1,3 Butanediol) 20 or 40 g will be ingested (open-label) before bedtime.

SUMMARY:
Obstructive Sleep Apnea (OSA) is a common medical disorder that is associated with reduced quality of life and higher risk of cardiovascular disease. Treatments for OSA and limited and not well tolerated. Our lab has shown that a low carbohydrate, high fat ketogenic diet (KD) can reduce OSA severity. Since it can be challenging to adhere to a ketogenic diet, the investigators propose that ingesting exogenous ketones can be an alternative method to improve OSA. Specifically the investigators will examine the effect of taking a commercially available product (Ketone-IQ) at bedtime on overnight ketones and sleep quality. The investigators will also examine the effect of Ketone-IQ on sleep apnea severity, compared to placebo.

This project will examine the pharmacokinetics, tolerability, and sleep impacts of ingesting exogenous ketones before sleep in patients with sleep apnea, while under treatment for OSA.

[Aim 2: Examine the preliminary efficacy of ingesting exogenous ketones before sleep on OSA]

DETAILED DESCRIPTION:
Sleep is a vulnerable period during which blunted respiratory drive and low airway muscle tone can cause dangerous breathing disorders. Obstructive sleep apnea (OSA) describes the intermittent collapse of the upper airway that induces O2 desaturations and arousals from sleep, placing patients at risk for cardiovascular disease, stroke, and death. In some obese patients, sleep causes carbon dioxide (CO2) accumulation progressing to daytime hypercapnia, a condition called obesity hypoventilation syndrome (OHS). Continuous positive airway pressure (CPAP) treats OSA and OHS, but is poorly tolerated, and may not fully correct sleep dysfunction.

Changes in metabolism may help to control OSA or OHS. The investigators recently published results from the Ketogenic Diet for OHS clinical trial (KETOHS, NCT04108819) showing that a 2-week ketogenic diet (high fat, low carbohydrate) for patients with OSA and OHS lowered reduced CO2, serum bicarbonate (HCO3), respiratory quotient, nocturnal hypoxemia(2). KD also significantly improved OSA. After participants resumed their prior diet, CO2 returned to baseline. The mechanisms by which KD improves sleep in this population could be related to reduced CO2 production (through fat oxidation), lowering of body weight, or direct effects of ketone bodies on sleep and breathing.

It is difficult to adhere long-term to KD, and there are multiple effects of this diet that make it challenging to understand mechanistic impacts on respiration. The investigators hypothesize that increasing ketone levels in the body, without having to adhere to a ketogenic diet, may be another method to improve breathing during sleep. Indeed, some drugs affecting acid-base status (e.g. acetazolamide or sulthiame) improve OSA, presumably through increasing and stabilizing respiratory drive. In this pilot study, the investigators will examine the pharmacokinetics, tolerability, and impacts of ingesting exogenous ketones (which are commercially available products) on sleep and breathing.

The specific ketone product to be tested for its impact on sleep and breathing is 1,3 butanediol (1,3BD) in a commercially available formulation called "Ketone IQ". 1,3BD is converted by liver metabolism into the ketone body beta-hydroxybutyrate (BHB) and has been utilized in multiple studies.

This project will be conducted in two studies, KETO-SLEEP 1 (KS1), and KETO-SLEEP 2 (KS2).

KETO-SLEEP 1: Examine the pharmacokinetics, tolerability, and sleep impacts of ingesting exogenous ketones (EK) before sleep (n=20, 10 men, 10 women). KS1 will lay the foundation for KS2 and other studies that administer exogenous ketones at bedtime, through dose-finding and assessment of tolerability. Patients with moderate-severe OSA (apnea-hypopnea index (AHI) >15)) adherent to CPAP will ingest EK or placebo 30 minutes before sleep. They will measure capillary BHB levels before ingestion and at 1, 3, 5, hours post-ingestion as well as upon awakening. CPAP use will be maintained on all nights and sleep architecture will be monitored with portable EEG. Questionnaires will solicit feedback about EK palatability, GI side effects, and sleep quality. Two doses (20 g and 40 g) of Ketone-IQ will be tested each for two nights, with one night used to measure BHB levels and separate night to allow for uninterrupted sleep.

[KETO-SLEEP 2: Examine the preliminary efficacy of ingesting exogenous ketones before sleep on OSA (n=20, 10 men, 10 women). KS2 will examine the respiratory effects of exogenous ketones taken before sleep. Patients with known OSA will be asked to temporarily discontinue CPAP, a technique used in our laboratory to temporarily elicit OSA(10). To account for night-to-night variability in OSA severity the investigators will use portable sleep monitoring to collect sleep and respiratory data two nights under each condition. The dose of Ketone-IQ to be administered each night will vary from 20 to 40 g, depending upon results of KS-1.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-65 years old with a BMI of 18 - 35 kg/m2
2. History of moderate-severe OSA as defined by AHI >15 events/hr (American Academy of Sleep Medicine criteria),
3. Adherent to CPAP (objectively determined via device download over last 30 days) using CPAP at least 70% of days for >=4 hours.
4. CPAP pressure ≤10 cm water (H2O) (based on prescribed CPAP pressure, or median pressure on an auto-titrating CPAP device).

Exclusion Criteria:

1. No concomitant sleep disorder (such as insomnia, restless leg syndrome, narcolepsy, idiopathic hypersomnia)
2. No current daytime respiratory impairment such as uncontrolled asthma, or uncontrolled chronic obstructive pulmonary disease (COPD), pneumonia, interstitial lung disease.
3. No use of supplemental oxygen.
4. Currently on a low carbohydrate (<130 g carbohydrate/day) or ketogenic diet, intermittent fasting, or consuming exogenous ketones
5. Pregnancy or breastfeeding
6. Alcohol consumption of > 10 standard drinks per week
7. Use of nightly medications that affect breathing (e.g. opiates, acetazolamide)
8. Use of Sodium-glucose cotransporter-2 (SGLT2) inhibitors. For example, Canagliflozin (Invokana), Dapagliflozin (Farxiga), Empagliflozin (Jardiance), Ertugliflozin (Steglatro)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Beta hydroxybutyrate (BHB) maximal concentration (Cmax) | Night 2, Night 5
  Participants will measure their capillary BHB levels at home at 4 time points after ingestion (1, 3, 5 hours, and final awakening). The investigators will derive the maximal BHB concentration (mmol) of these timepoints. Measured on two occasions: Night 2 (Ketone IQ 20 g) and Night 5 (Ketone IQ 40 g).

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Jun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Experimental data, including sleep data, questionnaires, and BHB measurements, will be stored as raw files on internal servers with cloud backup. Questionnaire data will be securely stored at Johns Hopkins University for three years post-study. Dr. Jun will control access to physical documents.
  Documentation and Accessibility: Research protocols, instrument details, and analysis methods will be detailed in publications. Deidentified data from published studies will be available at publication, accompanied by a data dictionary, and preserved for at least five years. Standard software (Excel, R, SPSS, SAS) will be used for data access and analysis.
Supporting Information: Study Protocol
Time Frame: Deidentified scientific data included in published manuscripts will be made available at the time of publication and additional data will be made available to researchers upon request. Data will be made available for up to 3 years following study completion.
Access Criteria: To request access to the data, researchers will be able to contact Dr. Jonathan Jun via email. Any data attached as a supplement to publications will be available for download from the publisher's website. The intention is to allow qualified external investigators broad access to the study data for specified research purposes.